CLINICAL TRIAL: NCT02704260
Title: Endofibrose Vasculaire et génétique
Brief Title: Genetic of SportS Induced Endofibrotic Remodeling
Acronym: GOSSER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A00441-48
Record Dates: First submitted 2016-02-23; First posted 2016-03-09 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2016-12

CONDITIONS: Genetic Syndrome
MeSH Terms: conditions — Genetic Diseases, Inborn | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GENETIC ANALISYS (Experimental): GENETIC ANALYSIS AND RESEARCH OF GENETIC BLOOD SAMPLE
  Interventions: Genetic: GENETIC ANALYSIS

INTERVENTIONS:
Genetic: GENETIC ANALYSIS — prélevement blood to search for a genetic cause of vascular endofibrose. Search genetic mutations in 5 subjects.

SUMMARY:
search for a genetic cause of vascular endofibrose

DETAILED DESCRIPTION:
Perform a DNA analysis to mark the existence of mutations in one or more genes encoding proteins involved in vascular remodeling high.

5 patients or relatives of patients topics

ELIGIBILITY:
Inclusion Criteria:

* High level reached Cyclists vascular endofibrose
* Cyclist high level and not sick with a brother or sister is senior cyclist reaches the vascular endofibrose.

Exclusion Criteria:

* not obtaining consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2016-09-02 (Actual); Study Completion 2016-09-02 (Actual)

PRIMARY OUTCOMES:
Presence of mutations or nucleotides variations | 1 hour
  DNA analysis and search for genetic mutations

CONTACTS AND LOCATIONS:
Overall Officials: PIERRE ABRAHAM, PROFESSOR, Principal Investigator — UH ANGERS
Locations (1):
- University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided